CLINICAL TRIAL: NCT01744275
Title: High Dose Omega 3 Fatty Acids Supplementation in Patients With Epilepsy : The HOPE-Epilepsy Trial
Brief Title: HOPE-Epilepsy Trial
Acronym: HOPE-Epilepsy
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCor; Research Institute - HCor (Other: HCor)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; Omega 3 fatty acids
MeSH Terms: conditions — Epilepsy | interventions — Fatty Acids, Omega-3; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: corn oil
- Omega 3 fatty acids supplementation (Experimental): Omega 3 fatty acids capsules
  Interventions: Dietary Supplement: Omega 3 fatty acids

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acids
  Arms: Omega 3 fatty acids supplementation
Dietary Supplement: corn oil — Placebo
  Arms: Placebo

SUMMARY:
This a multi-center study to examine whether supplementation with omega 3 fatty acids will reduce seizure frequency in patients with epilepsy .

ELIGIBILITY:
Inclusion Criteria:

* Patients with active Epilepsy

Exclusion Criteria:

* pregnant women or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Seizure Frequency | 18 months
  number of seizures during the treatment period

SECONDARY OUTCOMES:
categorized seizure frequency | 18 months
  number of crises categorized as: generalized, focal with disconnection and focal without disconnection
Percentage of overall seizure frequency modification | 18 months
  percentage of reduction or increase in seizure frequency from baseline til the end of treatment period
Time Free of seizures during treatment | 12 months
Reduction in seizure frequency | 12 months
Quality of Life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: M J Carrion, MD, Principal Investigator — Hospital do Coracao; O Berwanger, PhD, Study Chair — Hospital do Coracao; R D Lopes, PhD, Study Chair — BCRI; F A Scorza, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Research Institute, Hospital do Coração, São Paulo, São Paulo, Brazil